CLINICAL TRIAL: NCT01466595
Title: A Pilot Study of Rifaximin as a Modulator of Gut Microbial Translocation and Systemic Immune Activation in HIV-Infected Individuals With Incomplete CD4+ T-cell Recovery on Antiretroviral Therapy
Brief Title: Rifaximin as a Modulator of Microbial Translocation and Immune Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5286; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-10-06; First posted 2011-11-08 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Treatment with rifaximin (Experimental): Participants were administered one 550 mg tablet of rifaximin to be taken orally two times a day for 4 weeks.
  Interventions: Drug: Rifaximin
- Arm B: No study treatment (No Intervention): No study treatment for 4 weeks

INTERVENTIONS:
Drug: Rifaximin — Participant were administered one 550 mg tablet of rifaximin to be taken orally two times a day for 4 weeks.
  Arms: Arm A: Treatment with rifaximin

SUMMARY:
This study is being done to see whether rifaximin, an antibiotic that works in the intestines, can lower the amount of germs in the intestines of HIV infected persons. It is possible that when the amount of these germs is lowered, an HIV-infected person's immune system will become less active and will have a better chance of recovering. Also, the study will evaluate the safety of using rifaximin in HIV-infected subjects.

DETAILED DESCRIPTION:
A5286 is a randomized, open-label, two-arm, pilot (phase II) study that evaluated whether 4 weeks of treatment with rifaximin, a non-absorbable antibiotic, decreases markers of immune activation and levels of translocated gut microbial products in HIV-1 infected subjects virally suppressed on ART with CD4+ T-cells < 350 cells/mm^3. Rifaximin were admistered to subjects for 3 weeks. Follow-up continued to week 12. The total sample size was 73 subjects. Subjects were randomized at a 2:1 ratio (rifaximin: no study treatment), using permuted blocks, without institutional balancing.

Subjects were seen through week 12 for clinical and laboratory evaluations, including plasma HIV-1 RNA, CD4+ T-cell count, and safety laboratories. Subjects had 2 baseline visits -- at pre-entry and entry. Study visits were scheduled at weeks 2, 4, 8, and 12. CD4+ T-cell counts and HIV-1 RNA were measured at all weeks; measures of activations, gut-homing markers, and soluble biomarkers were also performed at all weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On ART for at least 96 weeks prior to study entry with a regimen that includes three or more antiretroviral medications. (Ritonavir ≤ 400 mg/day will not be considered a separate antiretroviral agent.)
* No plans to change the antiretroviral regimen at least in the next 3 months after study entry.
* CD4+ cell count < 350 cells/mm3 obtained within 120 days prior to study entry at any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
* All previous CD4+ cell counts should be < 350 cells/mm3 for at least 96 weeks prior to study entry while subjects were on ART. (A single CD4+ cell count ≥ 350 cells/mm3 is permitted within 96 weeks prior to study entry while subjects were on ART.)
* Documentation of HIV-1 RNA below the limit of detection (e.g., < 50 copies/mL on Roche Amplicor HIV-1 Monitor assay, < 75 copies/mL on the Versant HIV-1 RNA assay by branched DNA, < 400 copies/mL on a standard Roche Amplicor assay, < 40 copies/mL on the Abbott m2000sp/m2000rt real-time PCR test, < 48 copies/mL on the COBAS AmpliPrep/TAQMAN HIV-1 assay) verified by at least two measurements prior to study entry, one of which must be at least 48 weeks prior to study entry and one measurement that was obtained between 121 days and 48 weeks prior to study entry.
* Screening HIV-1 RNA below the limit of detection obtained within 120 days prior to study entry using a FDA -approved assay (e.g., < 50 copies/mL on Roche Amplicor HIV-1 Monitor assay, < 75 copies/mL on the Versant HIV-1 RNA assay by branched DNA, < 40 copies/mL on the Abbott m2000sp/m2000rt real-time PCR test, < 48 copies/mL on the COBAS AmpliPrep/TAQMAN HIV-1 assay). (The virologic assay must have a lower limit of detection of ≤ 75 copies/mL.)
* All other plasma HIV-1 RNA measurements in the 48 weeks prior to study entry must be below the limit of detection. (A single detectable measurement of ≤ 200 copies/mL is permitted if RNA levels immediately before and after are below the limits of detection for the assay.)
* Certain fasting laboratory values obtained within 45 days prior to entry as indicated in Section 4.1.9 of the protocol.
* Pre-entry peripheral blood mononuclear cell (PBMC) specimen for assay of the primary immune activation endpoint (change in CD8+ T-cells activation (%HLA-DR+CD38+CD8+ T-cells) has been obtained. Sites must receive confirmation from the processing lab via phone, e-mail, or fax, that this specimen has been entered into the ACTG's Laboratory Data Management System (LDMS).
* Female subjects of reproductive potential must have a negative serum or urine β-HCG pregnancy test with a sensitivity of at least 50 mIU/mL performed within 24 hours prior to study entry.
* If participating in sexual activity that could lead to pregnancy, the female subject must agree to use one form of contraceptive as listed in section 4.1.11 of the protocol while receiving protocol-specified treatment and for 4 weeks after stopping the treatment.
* If the female subject is not of reproductive potential, she is eligible without requiring the use of a contraceptive. Self report is acceptable documentation of sterilization, other contraceptive methods, and menopause.
* Ability and willingness of subject or legally authorized representative to provide informed consent.

Exclusion Criteria:

* Active diarrhea (3 or more unformed stools per day) within 28 days prior to study entry (except if site investigator or primary care provider attributes diarrhea to antiretroviral or azithromycin use).
* History of or active inflammatory bowel disease.
* History of or active Clostridium difficile colitis.
* History of significant liver disease, defined as having chronic liver disease (including chronic alcoholic liver disease, hepatitis B or C), plus either: a) ascites, b) encephalopathy, or c) a Child-Pugh Score of > 7.
* Receipt of antimicrobial therapy within 30 days prior to study entry. (NOTE: Antimicrobial use for prophylaxis of opportunistic infections, e.g., azithromycin or trimethoprim-sulfamethoxazole, is allowed.)
* Active infection requiring the use of antibiotics within 30 days prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study drug or their formulation (e.g., allergy to rifampin).
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to entry.
* Use of any of the following medications for more than 3 consecutive days within the 60 days prior to study entry:

  * Immunosuppressives
  * Immune modulators
  * Antineoplastic agents
  * Probiotics
  * Anticoagulants
* Vaccinations within 1 week prior to the pre-entry or study entry visits. (NOTE: Subjects are encouraged to get the flu vaccine prior to study pre-entry visit.)
* Participation on any HIV immunotherapy/therapeutic vaccination trials within 6 months prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan R. Tenorio, M.D., Study Chair — Rush University Medical Center
Locations (32):
- United States (31):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Stanford CRS (501), Palo Alto, California
  - Ucsf Aids Crs (801), San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS (103), Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS (31477), Newark, New Jersey
  - Cornell CRS (7804), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - HIV Prevention & Treatment CRS (30329), New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - Univ. of Rochester ACTG CRS (1101), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Derived] Tenorio AR, Chan ES, Bosch RJ, Macatangay BJ, Read SW, Yesmin S, Taiwo B, Margolis DM, Jacobson JM, Landay AL, Wilson CC; A5286 Team. Rifaximin has a marginal impact on microbial translocation, T-cell activation and inflammation in HIV-positive immune non-responders to antiretroviral therapy - ACTG A5286. J Infect Dis. 2015 Mar 1;211(5):780-90. doi: 10.1093/infdis/jiu515. Epub 2014 Sep 11. PMID 25214516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5286 opened under version 2.0 on 09/01/11, and the first subject was randomized on 10/03/11. Accrual to the study closed on 07/30/12, with a total of 73 subjects enrolled from 32 sites within the US.
Pre-assignment Details: Subjects were randomized with a 2:1 ratio (Rifaximin : no study treatment) at enrollment.
Period: Overall Study
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Started | 49 | 24
Completed | 49 | 23
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment | Total
Number analyzed (Participants) | 49 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 24 | 70
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.1) | 49.7 (9.7) | 49.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 45 | 22 | 67
Region of Enrollment [Number; unit: participants]
  United States | 49 | 24 | 73
Number of participants with HIV-1 RNA below assay lower limit [Number; unit: participants] — The number of participants with HIV-RNA below assay lower limit (<40 copies/mL) at baseline
  participants | 49 | 24 | 73
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — Total CD4+ T-cell count at baseline
  cells/mm^3 | 240 [197 to 284] | 223 [176 to 283] | 236 [189 to 284]

OUTCOME MEASURES:

1. Primary Outcome: Change in CD8+ T-cell Activation From Baseline to Week 4
Description: Change in CD8+ T-cell activation percent co-expressing HLA-DR and CD38 from baseline to week 4, where the baseline value is the average of pre-entry and entry values.
Time Frame: At baseline and 4 weeks
Population: The primary analysis is as-treated, limited to subjects who had data for both baseline and week 4, and (for the rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change antiretroviral therapy (ART) or use prohibited medications or have virologic failure during this time period.
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage HLA-DR+/CD38+ of CD8+ | 0.00 [-1.70 to 1.00] | 0.64 [0.11 to 1.48]
Statistical Analysis 1: Comparison: Arm A: Treatment With Rifaximin vs Arm B: No Study Treatment; Null hypothesis: There is no difference between the two arms in the change in T-cell activation from baseline to week 4; Test type: Superiority or Other; p = 0.028, Wilcoxon (Mann-Whitney) — not adjusted for multiple comparisons; no other adjustments

2. Secondary Outcome: Change in D-dimer From Baseline to Week 4
Description: Change in D-dimer from baseline to week 4, where baseline value is the average of pre-entry and entry.
  D-dimer is a fibrin degradation product (FDP), a small protein fragment present in the blood after a blood clot is degraded by fibrinolysis.
Time Frame: At baseline and 4 weeks
Population: This analysis is as-treated, limited to subjects who have data for baseline and week 4, and (for the Rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change ART or use prohibited medications or have virologic failure during this time period.
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | 0.00 [-0.12 to 0.06] | -0.03 [-0.14 to 0.04]

3. Secondary Outcome: Change in IL-6 From Baseline to Week 4
Description: Change in Interleukin (IL)-6 from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 pg/mL | -0.03 [-0.14 to 0.08] | 0.05 [-0.13 to 0.12]

4. Secondary Outcome: Change in LPS From Baseline to Week 4
Description: Change in Lipopolysaccharide (LPS) from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 pg/mL | 0.00 [-0.08 to 0.05] | -0.01 [-0.04 to 0.05]

5. Secondary Outcome: Change in hsCRP From Baseline to Week 4
Description: Change in High Sensitivity C-reactive Protein (Hs-CRP) from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | -0.08 [-0.29 to 0.15] | -0.09 [-0.21 to 0.16]

6. Secondary Outcome: Change in sCD14 From Baseline to Week 4
Description: Change in soluble CD14 (sCD14) from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | -0.03 [-0.07 to 0.06] | -0.03 [-0.05 to 0.01]

7. Secondary Outcome: Change in Peripheral B7hi CD4+ T-cell From Baseline to Week 4
Description: Change in gut-homing percent B7hi+ of CD4+ from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage B7hi+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage B7hi+ of CD4+ | -0.40 [-1.28 to 0.41] | 0.00 [-0.72 to 0.68]

8. Secondary Outcome: Change in %CD38+ of CD4+ From Baseline to Week 4
Description: Change in advanced flow percent CD38+ of CD4+ from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage CD38+ of CD4+ | 0.89 [-2.04 to 2.99] | 0.91 [-0.35 to 2.06]

9. Secondary Outcome: Change in %CD38+ of CD8+ From Baseline to Week 4
Description: Change in advanced flow percent CD38+ of CD8+ from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage CD38+ of CD8+ | 0.21 [-4.14 to 2.52] | 0.66 [0.18 to 3.03]

10. Secondary Outcome: Change in %Ki67+ of CD4+ From Baseline to Week 4
Description: Change in advanced flow percent Ki67+ of CD4+ from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage Ki67+ of CD4+ | -0.17 [-0.47 to 0.25] | 0.05 [-0.36 to 0.51]

11. Secondary Outcome: Change in %Ki67+ of CD8+ From Baseline to Week 4
Description: Change in advanced flow percent Ki67+ of CD8+ from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage Ki67+ of CD8+ | -0.12 [-0.27 to 0.12] | 0.12 [-0.07 to 0.27]

12. Secondary Outcome: Change in %HLA-DR+/CD38+ of CD4+ From Baseline to Week 4
Description: Change in CD4 activation percent co-expressing HLA-DR and CD38 from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
percentage HLA-DR+/CD38+ of CD4+ | -0.15 [-1.03 to 0.99] | 0.15 [-0.59 to 0.86]

13. Secondary Outcome: Change in CD38+ of CD8+ MFI From Baseline to Week 4
Description: Change in CD38+ of CD8+ MFI (Median Fluorescence Intensity) from baseline to week 4, where baseline value is the average of pre-entry and entry.
  MFI measures the shift in fluorescence intensity of a population of cells. MFI values are based on control to demonstrate an increase or decrease in expression of the marker. MFI in this study was automatically calculated in FlowJo. The median is the relative intensity value below which 50% of the events are found. MFI is an arbitrary unit of relative intensity.
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: MFI (relative intensity)
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
MFI (relative intensity) | 0.00 [-0.04 to 0.07] | 0.03 [0.00 to 0.07]

14. Secondary Outcome: Change in CD4 Count From Baseline to Week 4
Description: Change in total CD4 T-cell from baseline to week 4, where baseline value is the average of pre-entry and entry
Time Frame: At baseline and 4 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
cells/mm3 | -3.00 [-20.50 to 31.00] | 11.25 [-9.00 to 52.00]

15. Secondary Outcome: Change in CD8+ T-cell Activation From Week 4 to Week 8
Description: Change in CD8+ T-cell activation percent co-expressing HLA-DR and CD38 from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: This analysis is as-treated, limited to subjects who had data for both week 4 and week 8, and (for the rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change ART or use prohibited medications or have virologic failure prior to week 8.
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage HLA-DR+/CD38+ of CD8+ | 0.08 [-0.70 to 0.70] | -0.71 [-1.85 to 0.56]

16. Secondary Outcome: Change in D-dimer From Week 4 to Week 8
Description: D-dimer is a fibrin degradation product (FDP), a small protein fragment present in the blood after a blood clot is degraded by fibrinolysis.
Time Frame: At weeks 4 and 8
Population: This analysis is as-treated, limited to subjects who have data for week 4 and week 8, and (for the Rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change ART or use prohibited medications or have virologic failure prior to week 8
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
log10 ng/mL | -0.02 [-0.10 to 0.09] | 0.03 [-0.03 to 0.17]

17. Secondary Outcome: Change in IL-6 From Week 4 to Week 8
Description: Change in IL-6 from week 4 to week 8.
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
log10 pg/mL | -0.03 [-0.18 to 0.08] | 0.06 [-0.01 to 0.19]

18. Secondary Outcome: Change in LPS From Week 4 to Week 8
Description: Change in LPS from week 4 to week 8.
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
log10 pg/mL | -0.01 [-0.08 to 0.02] | 0.00 [-0.03 to 0.07]

19. Secondary Outcome: Change in hsCRP From Week 4 to Week 8
Description: Change in hsCRP from week 4 to week 8.
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
log10 ng/mL | -0.05 [-0.29 to 0.20] | 0.23 [0.06 to 0.50]

20. Secondary Outcome: Change in sCD14 From Week 4 to Week 8
Description: Change in soluble CD14 from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
log10 ng/mL | -0.05 [-0.11 to 0.04] | 0.02 [-0.03 to 0.05]

21. Secondary Outcome: Change in Peripheral B7hi CD4+ T-cells From Week 4 to Week 8
Description: Change in gut homing percent B7hi+ of CD4+ from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage B7hi+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage B7hi+ of CD4+ | 0.26 [-0.37 to 0.97] | -0.02 [-0.82 to 1.06]

22. Secondary Outcome: Change in %CD38+ of CD4+ From Week 4 to Week 8
Description: Change in advanced flow percent CD38+ of CD4+ from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage CD38+ of CD4+ | -0.84 [-3.2 to 1.33] | 1.00 [-1.88 to 2.92]

23. Secondary Outcome: Change in %CD38+ of CD8+ From Week 4 to Week 8
Description: Change in advanced flow percent CD38+ of CD8+ from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage CD38+ of CD8+ | -0.12 [-2.30 to 2.09] | -1.20 [-3.04 to 1.84]

24. Secondary Outcome: Change in %Ki67+ of CD4+ From Week 4 to Week 8
Description: Change in advanced flow percent Ki67+ of CD4+ from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage Ki67+ of CD4+ | 0.21 [-0.17 to 0.53] | -0.01 [-0.58 to 0.51]

25. Secondary Outcome: Change in %Ki67+ of CD8+ From Week 4 to Week 8
Description: Change in advanced flow percent Ki67+ of CD8+ from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage Ki67+ of CD8+ | 0.11 [-0.05 to 0.23] | -0.08 [-0.21 to 0.06]

26. Secondary Outcome: Change in CD4 Activation Percent From Week 4 to Week 8
Description: Change in CD4 activation percent co-expressing HLA-DR and CD38 from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
percentage HLA-DR+/CD38+ of CD4+ | 0.17 [-0.66 to 0.86] | -0.53 [-0.85 to 0.31]

27. Secondary Outcome: Change in CD38+ of CD8+ MFI From Week 4 to Week 8
Description: Change in CD38+ of CD8+ median fluorescence intensity (MFI) from week 4 to week 8.
  MFI measures the shift in fluorescence intensity of a population of cells. MFI values are based on control to demonstrate an increase or decrease in expression of the marker. MFI in this study was automatically calculated in FlowJo. The median is the relative intensity value below which 50% of the events are found. MFI is an arbitrary unit of relative intensity.
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: MFI (relative intensity)
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 21
MFI (relative intensity) | 0.08 [-0.70 to 0.70] | -0.71 [-1.85 to 0.56]

28. Secondary Outcome: Change in CD4 Count From Week 4 to Week 8
Description: Change in total CD4 T-cell count from week 4 to week 8
Time Frame: At weeks 4 and 8
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 21
cells/mm3 | -9.50 [-26.00 to 9.00] | -13.00 [-30.00 to 5.00]

29. Secondary Outcome: Change in CD8+ T-cell Activation From Week 4 to Week 12
Description: Change in CD8+ T-cell activation percent co-expressing HLA-DR and CD38 from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: This analysis is as-treated, limited to subjects who had data for both week 4 and week 12, and (for the rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change ART or use prohibited medications or have virologic failure prior to week 12.
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage HLA-DR+/CD38+ of CD8+ | -0.05 [-0.76 to 1.00] | -0.77 [-2.91 to 0.23]

30. Secondary Outcome: Change in D-dimer From Week 4 to Week 12
Description: as for outcome 16
Time Frame: At weeks 4 and 12
Population: This analysis is as-treated, limited to subjects who have data for week 4 and week 12, and (for the Rifaximin arm) remain on study treatment through week 4 (allowing less than or equal to 6 missed doses), and did not change ART or use prohibited medications or have virologic failure prior to week 12.
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | -0.01 [-0.10 to 0.09] | 0.07 [-0.02 to 0.10]

31. Secondary Outcome: Change in IL-6 From Week 4 to Week 12
Description: Change in IL-6 from week 4 to week 12.
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 pg/mL | 0.02 [-0.13 to 0.25] | 0.02 [-0.21 to 0.15]

32. Secondary Outcome: Change in LPS From Week 4 to Week 12
Description: Change in LPS from week 4 to week 12.
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 pg/mL | 0.00 [-0.09 to 0.04] | 0.03 [-0.01 to 0.12]

33. Secondary Outcome: Change in hsCRP From Week 4 to Week 12
Description: Change in hsCRP from week 4 to week 12.
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | 0.09 [-0.13 to 0.28] | 0.04 [-0.08 to 0.27]

34. Secondary Outcome: Change in sCD14 From Week 4 to Week 12
Description: Change in soluble CD14 from week 4 to week 12
Time Frame: At weeks 4 and 8
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 43 | 22
log10 ng/mL | 0.03 [-0.03 to 0.08] | 0.02 [-0.05 to 0.10]

35. Secondary Outcome: Change in Peripheral B7hi CD4+ T-cells From Week 4 to Week 12
Description: Change in gut homing percent B7hi+ of CD4+ from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage B7hi+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 41 | 22
percentage B7hi+ of CD4+ | -0.07 [-0.57 to 0.69] | -0.19 [-0.98 to 0.11]

36. Secondary Outcome: Change in %CD38+ of CD4+ From Week 4 to Week 12
Description: Change in advanced flow percent CD38+ of CD4+ from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage CD38+ of CD4+ | -0.67 [-3.81 to 2.91] | -0.54 [-4.82 to 1.81]

37. Secondary Outcome: Change in %CD38+ of CD8+ From Week 4 to Week 12
Description: Change in advanced flow percent CD38+ of CD8+ from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage CD38+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage CD38+ of CD8+ | -0.93 [-3.60 to 2.40] | -1.96 [-6.50 to 0.60]

38. Secondary Outcome: Change in %Ki67+ of CD4+ From Week 4 to Week 12
Description: Change in advanced flow percent Ki67+ of CD4+ from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage Ki67+ of CD4+ | 0.14 [-0.23 to 0.79] | -0.22 [-0.85 to 0.32]

39. Secondary Outcome: Change in %Ki67+ of CD8+ From Week 4 to Week 12
Description: Change in advanced flow percent Ki67+ of CD8+ from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage Ki67+ of CD8+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage Ki67+ of CD8+ | 0.13 [-0.11 to 0.37] | -0.09 [-0.16 to 0.16]

40. Secondary Outcome: Change in CD4 Activation Percent From Week 4 to Week 12
Description: Change in CD4 activation percent co-expressing HLA-DR and CD38 from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: percentage HLA-DR+/CD38+ of CD4+
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
percentage HLA-DR+/CD38+ of CD4+ | -0.14 [-0.70 to 1.03] | -0.50 [-1.65 to 0.16]

41. Secondary Outcome: Change in CD38+ of CD8+ MFI From Week 4 to Week 12
Description: Change in CD38+ of CD8+ median fluorescence intensity (MFI) from week 4 to week 12.
  MFI measures the shift in fluorescence intensity of a population of cells. MFI values are based on control to demonstrate an increase or decrease in expression of the marker. MFI in this study was automatically calculated in FlowJo. The median is the relative intensity value below which 50% of the events are found. MFI is an arbitrary unit of relative intensity.
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: MFI (relative intensity)
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
MFI (relative intensity) | -0.02 [-0.06 to 0.04] | -0.02 [-0.09 to 0.03]

42. Secondary Outcome: Change in CD4 Count From Week 4 to Week 12
Description: Change in total CD4 T-cell count from week 4 to week 12
Time Frame: At weeks 4 and 12
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 42 | 22
cells/mm3 | 0.00 [-26.00 to 20.00] | -5.50 [-44 to 39]

43. Secondary Outcome: Primary Adverse Events
Description: Primary adverse events include all SAEs, defined according to ICH guidelines and targeted protocol events (grade 2 or higher signs and symptoms, grade 2 or higher laboratory abnormality, all diagnoses identified by the ACTG criteria for clinical events, and all events that led to a change in treatment regardless of grade).
Time Frame: from study enrollment until study completion at 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Number analyzed (Participants) | 49 | 24
participants | 27 | 9

ADVERSE EVENTS:
Time Frame: AEs reported from study enrollment until study completion at 12 weeks
Description: AE reporting followed DAIDS Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and ≥grade 3 AEs (where grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death).
Arm/Group | Arm A: Treatment With Rifaximin | Arm B: No Study Treatment
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/24
Other Adverse Events (participants affected / at risk) | 36/49 | 19/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Treatment With Rifaximin (N=49) | Arm B: No Study Treatment (N=24)
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 4 | 1
Pyrexia (General disorders) | 3 | 1
Blood bilirubin increased (Investigations) | 7 | 2
Blood cholesterol increased (Investigations) | 18 | 12
Blood creatinine increased (Investigations) | 2 | 2
Blood glucose increased (Investigations) | 7 | 5
Blood phosphorus decreased (Investigations) | 2 | 3
Blood sodium decreased (Investigations) | 4 | 2
Blood uric acid increased (Investigations) | 1 | 4
Lipase abnormal (Investigations) | 0 | 2
Lipase increased (Investigations) | 2 | 2
Low density lipoprotein increased (Investigations) | 11 | 9
Neutrophil count decreased (Investigations) | 6 | 0
Platelet count decreased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Headache (Nervous system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No